CLINICAL TRIAL: NCT02248402
Title: A Phase 1/2a Study to Evaluate Safety and Efficacy of Autologous Dendritic Cell Therapy in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Autologous Dendritic Cell Therapy in Patients With Relapsed or Refractory Multiple Myeloma
Acronym: Vax-DC/MM
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Sung-Hoon Jung, M.D, Chonnam National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-038
Record Dates: First submitted 2014-09-17; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vax-DC/MM (Experimental)
  Interventions: Biological: Vax-DC/MM

INTERVENTIONS:
Biological: Vax-DC/MM

SUMMARY:
Multiple myeloma remains incurable disease in most patients . Cellular immunotherapy using dendritic cells is emerging as a useful immunotherapeutic modality to treat multiple myeloma. Vax-DC/MM is an potent immunotherapeutic agent generated by dendritic cells loaded with the ultraviolet B-irradiated autologous human myeloma cells. The main purpose of this study is to examine the safety and efficacy of Vax-DC/MM in patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
* To create the Vax-DC/MM, myeloma cells will be obtained from the bone marrow of the participants, and leukapheresis will be performed to obtain dendritic cells
* Not everyone who participants in this study will be receiving the same dose of study vaccine. A small group of patients will be enrolled into the study and given a certain dose. If they tolerate it, the next group of patients enrolled will received a higher dose.
* Before the first injection of Vax-DC, low dose cyclophosphamide will be administered to stimulate immune response.
* Participants will be received a certain dose of Vax-DC weekly four times.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory multiple myeloma who received at least one prior therapy including thalidomide, bortezomib, or lenalidomide-containing regimen
* Subjects with measurable disease defined as at least one of the following Serum M-protein ≥ 1.0 g/dL Urine M-protein ≥ 400 mg/24hr
* Eastern Cooperative Oncology Group Performance Status ≤ 2
* Hemoglobin ≥ 8 g/dL (≥ 4.96 mol/L): Prior red blood cell transfusion or recombinant human erythropoietin use is allowed.
* Absolute neutrophil count (ANC) ≥ 1.0 x 109/L
* Aspartate aminotransferase (AST) < 3 times the upper limit of normal
* Alanine aminotransferase (ALT) < 3 times the upper limit of normal
* Subjects (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Smoldering or indolent myeloma
* Uncontrolled or severe cardiovascular disease (cardiac ejection fraction<0.5, Severe conduction disorder )
* Sepsis or current active infection
* Pregnancy or breastfeeding
* Received other immunotherapy treatment
* Clinically significant autoimmune disease
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 1 years
  Adverse events were assessed using the National Cancer Institute common toxicity criteria (NCI-CTC) for adverse events version 4.0 every injection of Vax-DC/MM

SECONDARY OUTCOMES:
Clinical response after completion of Vax-DC/MM injection | 2 year
  The International Myeloma Working Group uniform criteria were used to assess the clinical response.
Progression free survival | 2 year
  Progression free survival was defined as the period from the start of treatment until the end follow-up or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Chonnam National University Hwasun Hospital, Hwasun, Jeollanamdo, South Korea